CLINICAL TRIAL: NCT05717829
Title: Modified Hip Capsular Incision: an Easier Way to do Hip Capsulorrhaphy in Developmental Dysplasia of the Hip (DDH)
Acronym: DDH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCIDDH
Record Dates: First submitted 2023-01-14; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Developmental Hip Dysplasia
Keywords: DDH; Developmental hip dysplasia; Capsulorrhaphy
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Intervention Model Description: prospective case series study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified hip capsular incision (Experimental): make re -suturing of the capsule easier with multiple stitches.
  Interventions: Procedure: Modified hip capsular incision

INTERVENTIONS:
Procedure: Modified hip capsular incision — modified incision to make re -suturing of the capsule easier with multiple stitches.

SUMMARY:
Developmental dysplasia of the hip (DDH) is the commonest hip problem seen by pediatric orthopaedic surgeons (1). DDH refers to an abnormal configuration of, or relationship between, the femoral head and the acetabulum .Principals of surgical treatment of DDH, however, always include reduction and stabilization. These principals could be applied by conservative or surgical means (2). Goal of Treatment options to Obtain and maintain reduction without damaging femoral head. Surgical Stabilization might be required in cases with failed conservative treatment, residual dysplasia or older children with neglected DDH. Surgical stabilization is generally achieved by a reduction into a near anatomical position and a complementary capsulorrhaphy (3). In the classic T-shaped capsular incision, the vertical branch parallel to the axis of the neck and the horizontal branch 5 mm from the iliac insertion of the capsule, from anterior and downward to posterior and upward. Two flaps are thus obtained (4). It was noticed that doing capsulorrhaphy after head reduction is cumbersome with this technique because it needs shallow-curved needles while suturing in narrow field and sometimes the suture material gets avulsed from medial flab. A suggested technique by doing a modified incision to make re -suturing of the capsule easier with multiple stitches.

DETAILED DESCRIPTION:
This Modified incision to make re -suturing of the capsule easier with multiple stitches.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-7 years old
* Primary DDH

Exclusion Criteria:

* Paralytic hip DX in cases of (Cerebral palsy,Meningomyelocele,Neuropathy or Myopathy)
* Recurrent cases of DDH

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of hip capsulorrhaphy | intraoperative
  as regards operative time to do capsullorrhapy in minutes

SECONDARY OUTCOMES:
Any complications detected | 1 year
  as: infection -Recurrent dislocation -AVN

CONTACTS AND LOCATIONS:
Overall Officials: Hesaham Elbaseet, MD, Principal Investigator — Assiut University
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves C, Truong WH, Thompson MV, Suryavanshi JR, Penny CL, Do HT, Dodwell ER. Diagnostic and treatment preferences for developmental dysplasia of the hip: a survey of EPOS and POSNA members. J Child Orthop. 2018 Jun 1;12(3):236-244. doi: 10.1302/1863-2548.12.180034. PMID 29951123
- [Background] Qadir I, Ahmad S, Zaman AU, Khan CM, Ahmad S, Aziz A. One-stage Hip Reconstruction for Developmental Hip Dysplasia in Children over 8 Years of Age. Hip Pelvis. 2018 Dec;30(4):260-268. doi: 10.5371/hp.2018.30.4.260. Epub 2018 Dec 6. PMID 30534545
- [Background] Glorion C. Surgical reduction of congenital hip dislocation. Orthop Traumatol Surg Res. 2018 Feb;104(1S):S147-S157. doi: 10.1016/j.otsr.2017.04.021. Epub 2017 Dec 2. PMID 29203431
- [Result] Clinical practice guideline: early detection of developmental dysplasia of the hip. Committee on Quality Improvement, Subcommittee on Developmental Dysplasia of the Hip. American Academy of Pediatrics. Pediatrics. 2000 Apr;105(4 Pt 1):896-905. doi: 10.1542/peds.105.4.896. PMID 10742345